CLINICAL TRIAL: NCT04678453
Title: Single Center, Open Label, Phase 1 Study to Evaluate the Safety, Tolerability and Exploratory Efficacy of SNK01 in Subjects With Alzheimer's Disease (AD)
Brief Title: Safety of SNK01 in Subjects With Alzheimer's Disease (ASK-AD)
Acronym: ASK-AD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated after completing the dose escalation portion of the study. The expansion cohort was not initiated to conduct a global trial based on the approved US IND using a new manufacturing process.
Sponsor: NKGen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNK01-MX04
Record Dates: First submitted 2020-12-09; First posted 2020-12-22 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease; Neuro-Degenerative Disease
Keywords: Natural killer cell; NK cell; Expanded natural killer cell; Alzheimer's Disease; Neurodegenerative diseases; Neurocognitive disorders; Brain diseases; Autologous natural killer cell
MeSH Terms: conditions — Alzheimer Disease; Neurodegenerative Diseases; Neurocognitive Disorders; Brain Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1 - Low dose SNK01 (Experimental): SNK01 (low dose) administered once every three weeks (Q3W) for four cycles.
  Interventions: Biological: SNK01
- Cohort 2 - Medium dose SNK01 (Experimental): SNK01 (medium dose) administered Q3W for four cycles.
  Interventions: Biological: SNK01
- Cohort 3 - High dose SNK01 (Experimental): SNK01 (high dose) administered Q3W for four cycles.
  Interventions: Biological: SNK01
- Cohort 4 - SNK01 at Maximum Tolerated Dose (MTD) / Recommended Phase 2 Dose (RP2D) (Experimental): SNK01 (at MTD/RP2D) administered Q3W for four cycles.
  Interventions: Biological: SNK01

INTERVENTIONS:
Biological: SNK01 — Patient-specific ex vivo expanded autologous natural killer cells

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary efficacy of SNK01 (autologous natural killer cell), as a single agent, for the treatment of subjects with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and protocol. If the subject is incapable of giving or signing informed consent, the subject must have a legally authorized representative willing to consent on their behalf.
* Subject must be ≥ 55 to 85 years old at the time of consent.
* Magnetic resonance imaging (MRI) scans of the brain within the past six months reveal evidence and findings consistent with Alzheimer's disease, including hippocampal volume loss and/or overall cerebral atrophy (cerebral volume loss).
* Fluorodeoxyglucose-positron emission tomography (FDG-PET) scans of the brain within the past six months reveal evidence and findings consistent with mild cognitive impairment or Alzheimer's disease.
* Subject presenting, during evaluation by the study Investigator, to have spontaneous memory loss or presenting abnormal memory function in early screening.
* Subject must be in good health with adequate hearing and vision.
* Subject must have a reliable caregiver.
* Women of childbearing potential who are not abstinent and intend to be sexually active with a nonsterilized male partner must be willing to use an adequate method of contraception throughout the study and for one month following the last day of the last administration of final study drug dose. Acceptable methods include hormonal contraception (oral contraceptives [taken 90 days prior to administration of study drug], intrauterine devices (IUD), or double barrier methods (e.g., vaginal diaphragm/vaginal sponge plus condoms, or condom plus spermicidal jelly), sexual abstinence, or a vasectomized partner.

Exclusion Criteria:

* Any medical or neurological conditions, other than Alzheimer's disease, that could contribute to the cause of cognitive impairment in the subject. Examples include, but are not limited to, frontotemporal dementia (FTD), Lewy body dementia, vascular dementia, Parkinson's disease, corticobasal degeneration, Creutzfeldt-Jakob disease, progressive supranuclear palsy, Huntington's disease, normal pressure hydrocephalus, seizure disorders or cerebral hypoxia, post-traumatic stress disorder (PTSD), or alcohol or medication use or abuse.
* Subject does not present with signs of mild cognitive impairment or Alzheimer's disease at screening, or during evaluation by the study Investigator.
* Subject presents with significant brain disease including hemorrhage or infarction.
* Subject has a history of cerebrovascular accident or transient ischemic attack (TIA), or unexplainable loss of consciousness during the past year.
* Subject has a history of schizophrenia, schizoaffective disorder, major depressive disorder (MDD), bipolar disorder, or any other clinically relevant psychiatric disease.
* Subject has a history of seizure episodes within the past three years.
* Subject has uncontrolled diabetes mellitus.
* Subject has a history of unstable angina, myocardial infarction, chronic heart failure, or clinically relevant conduction abnormalities within the year prior to screening.
* Subject suffers from renal or hepatic failure.
* Subject is infected with the human immunodeficiency virus (HIV), Hepatitis B (Hep B), Hepatitis C (Hep C), or any other infection or active systemic disease.
* Subject is using anticoagulants (except aspirin at or below a prophylactic dose).
* Subject is currently exceeding the normal recommended dosage for any drug used to treat Alzheimer's disease (e.g., memantine or acetylcholinesterase inhibitors [AChEI]).
* Subject has contraindication to MRI scans, FDG-PET scans, or lumbar spinal taps.
* Subject whose safety is considered to be at risk from trial's intervention, as determined by the study Investigator.
* Pregnant or lactating female subjects.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
To determine the safety profile of SNK01 monotherapy in patients with mild cognitive impairment (MCI) or Alzheimer's Disease by monitoring for adverse events. | Up to 6 months
  Evaluated by the number of treatment emergent adverse event (TEAE) Grade 3 or higher considered to be related to SNK01, adverse events (AEs) of Grade 3 or higher using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v5.0, measurements of vital signs, clinical laboratory tests and physical examination.
To determine the tolerability of SNK01 monotherapy in patients with mild cognitive impairment (MCI) or Alzheimer's Disease by monitoring for adverse events. | Up to 6 months
  Evaluated by the number of treatment emergent adverse event (TEAE) Grade 3 or higher considered to be related to SNK01, adverse events (AEs) of Grade 3 or higher using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v5.0, measurements of vital signs, clinical laboratory tests and physical examination.
To determine the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of SNK01 monotherapy. | Up to 6 months
  Assessed by the incidence of dose-limiting toxicities, defined by treatment emergent adverse event (TEAE) Grade 3 or higher considered to be related to SNK01, in each dose level.

SECONDARY OUTCOMES:
To assess preliminary efficacy of SNK01 measured by Alzheimer's Disease Assessment Scale Cognitive subscale (ADAS-Cog). | Baseline, Week 11, End of Study (Week 22)
To assess preliminary efficacy of SNK01 measured by Mini-Mental Status Exam (MMSE). | Baseline, Week 11, End of Study (Week 22)
To assess preliminary efficacy of SNK01 measured by Clinical Dementia Rating Scale: Sum of Boxes (CDR-SB). | Baseline, Week 11, End of Study (Week 22)
To assess preliminary efficacy of SNK01 measured by Alzheimer's Disease Composite Score (ADCOMS). | Baseline, Week 11, End of Study (Week 22)
To assess preliminary efficacy of SNK01 measured by cerebrospinal fluid (CSF) biomarkers: amyloid beta 42, T-tau and P-tau. | Baseline, Week 11, End of Study (Week 22)

CONTACTS AND LOCATIONS:
Overall Officials: Clemente Humberto Zúñiga Gil, MD, Principal Investigator — Hospital Angeles Tijuana
Locations (1):
- Hospital Angeles Tijuana, Tijuana, Estado de Baja California, Mexico

REFERENCES:
- [Derived] Zuniga CH, Acosta BI, Menchaca R, Amescua CA, Hong S, Hui L, Gil M, Rhee YH, Yoon S, Kim M, Chang PY, Kim YM, Song PY, Betito K. Treatment of Alzheimer's Disease subjects with expanded non-genetically modified autologous natural killer cells (SNK01): a phase I study. Alzheimers Res Ther. 2025 Feb 12;17(1):40. doi: 10.1186/s13195-025-01681-2. PMID 39939891